CLINICAL TRIAL: NCT02195011
Title: A Two Arm Safety Study of Regorafenib Before or After SIR-Spheres Microspheres (90Y) for the Treatment of Patients With Refractory Metastatic Colorectal Cancer With Liver Metastases
Brief Title: Safety Study of Regorafenib and SIR-Spheres® Microspheres Radioembolization in Patients With Refractory Metastatic Colorectal Cancer With Liver Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Sirtex Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GI 189
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms
Keywords: Regorafenib; 90Y; Radioembolization; SIR-Spheres Microspheres; Metastatic Colorectal Cancer; Liver Metastases; SIRT; Refractory
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Cohort 1: Regorafenib/SIR-Spheres/Regorafenib (Experimental): Regorafenib (one cycle) followed by SIR-Spheres followed by re-initiation of regorafenib 2-4 weeks after SIR-Spheres.
  Patients will take regorafenib 160 mg orally once daily on Days 1-21 of each 28-day treatment cycle. SIR-Spheres microspheres will then be administered to the patient by injection through a trans-femoral catheter into the hepatic artery. Treatment with regorafenib will be re-started 2-4 weeks after SIR-Spheres administration.
  Interventions: Device: SIR-Spheres; Drug: Regorafenib
- Cohort 2: SIR-Spheres/Regorafenib (Experimental): SIR-Spheres followed by regorafenib to start 2-4 weeks after SIR-Spheres.
  SIR-Spheres microspheres will be administered to the patient by injection through a trans-femoral catheter into the hepatic artery. After SIR-Spheres microspheres have been administered, the treatment with regorafenib will be initiated 2-4 weeks after administration of SIR-Spheres. Patients will take regorafenib 160 mg orally once daily on Days 1-21 of each 28-day treatment cycle.
  Interventions: Device: SIR-Spheres; Drug: Regorafenib

INTERVENTIONS:
Device: SIR-Spheres — Radioembolization will be administered once by injection through a trans-femoral catheter into the hepatic artery.
  Other Names: 90Y-Microspheres
Drug: Regorafenib — All patients will take regorafenib 160mg orally once daily on Days 1-21 of each 28-day cycle.
  Other Names: Stivarga

SUMMARY:
The purpose of this study is to determine the safety of regorafenib, an antiangiogenic drug, when combined with radioembolization using SIR-Spheres® microspheres in the treatment of colorectal cancer (CRC) that has spread to the liver.

DETAILED DESCRIPTION:
Recent targeted therapies and treatment strategies have shown promise in colorectal cancer; however, elimination of disease remains a challenge once spread to the liver. Radioembolization using SIR-Spheres® microspheres (SIR-Spheres) to treat liver-only or liver-dominant metastatic colorectal cancer (mCRC) has been successful in this refractory setting. In this open-label study we will compare the safety of two treatment cohorts in which radioembolization will be administered using the device SIR-Spheres microspheres (90Y resin microspheres) in combination with regorafenib to patients with mCRC with liver metastases. The two treatment cohorts will be evaluated for safety, overall response (OR), progression-free survival (PFS), and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic adenocarcinoma of the colon or rectum.
2. Patients who have been previously treated with or are not candidates for fluorouracil, oxaliplatin, irinotecan, and if Kras wild-type, anti EGFR therapy.
3. Considered an appropriate candidate for regorafenib therapy.
4. Measurable disease or evaluable disease as measured by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Measurable computed tomography (CT) scan evidence of liver metastases which are not treatable by surgical resection or local ablation with curative intent at the time of study entry.
6. ECOG Performance Status score of 0-1.
7. Adequate hematologic, renal and liver function.
8. Male patients with female partners of childbearing potential and women female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 30 days following last dose.
9. Life expectancy ≥ 3 months.
10. Ability to understand the nature of this study and give written informed consent

Exclusion Criteria:

1. Most recent chemotherapy ≤14 days and ≥Grade 1 chemotherapy-related side effects, with the exception of alopecia.
2. Use of a study drug ≤21 days or 5 half-lives (whichever is shorter) prior to initiation of study treatment. For study drugs for which 5 half-lives is ≤21 days, a minimum of 10 days between termination of the study drug and administration of study treatment is required.
3. Wide field radiotherapy (including therapeutic radioisotopes such as strontium-89 administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
4. Previous radiation delivered to the upper abdomen.
5. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
6. Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 2 weeks previously and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
7. Leptomeningeal metastases or spinal cord compression due to disease.
8. Pregnant or lactating.
9. Evidence of ascites, cirrhosis, portal hypertension, or thrombosis as determined by clinical or radiologic assessment.
10. History of abdominal fistula or gastrointestinal perforation ≤6 months prior to beginning study treatment.
11. Serious non-healing wound, active ulcer, or untreated bone fracture.
12. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (e.g. ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, and malabsorption syndrome).
13. Any of the following cardiac diseases currently or within the last 6 months:

    * Unstable angina pectoris
    * Congestive heart failure (NYHA ≥ Grade 2)
    * Conduction abnormality not controlled with pacemaker or medication
    * Significant ventricular or supraventricular arrhythmias (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
    * Valvular disease with significant compromise in cardiac function
14. Inadequately controlled hypertension (i.e., systolic blood pressure [SBP] >180 mmHg or diastolic blood pressure (DBP) >100 mmHg) (patients with values above these levels must have their blood pressure (BP) controlled with medication prior to starting treatment).
15. Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
16. Known diagnosis of human immunodeficiency virus, hepatitis B, or hepatitis C.
17. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
18. Use of strong CYP34A inducers or inhibitors.
19. The herbal medications St. John's wort, kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng will not be allowed during study treatment. Patients should stop using these herbal medications 7 days prior to first dose of study drug.
20. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
21. Inability or unwillingness to comply with study and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-06-04 (Actual); Study Completion 2017-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Kennedy, MD, Study Chair — SCRI Development Innovations, LLC; Johanna Bendell, MD, Study Chair — SCRI Development Innovations, LLC
Locations (3):
- United States (3):
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Research Medical Center, Kansas City, Missouri
  - Tennessee Oncology PLLC, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between July 2014 and February 2017, 26 patients with metastatic colorectal cancer (mCRC) with liver metastases were enrolled. The study was closed early due to slow enrollment.
Groups:
- Cohort 1: Regorafenib/SIR-Spheres/Regorafenib: Patients with metastatic colorectal cancer (mCRC) with liver metastases received one cycle (28 days) of regorafenib followed by SIR-Spheres followed by re-initiation of regorafenib 2-4 weeks after SIR-Spheres.
  Patients in Cohort 1 took 160 mg regorafenib orally once daily on Days 1-21 of each 28-day treatment cycle. SIR-Spheres microspheres were then be administered to patients by injection via trans-femoral catheter into the hepatic artery. Following treatment with SIR-Spheres, patients took 160 mg regorafenib orally once daily on Days 1-21 of each 28-day treatment cycle
- Cohort 2: SIR-Spheres/Regorafenib: Patients with metastatic colorectal cancer (mCRC) with liver metastases received SIR-Spheres microspheres followed by regorafenib to start 2-4 weeks after SIR-Spheres.
  Patients in Cohort 2 received SIR-Spheres microspheres administered by injection via trans-femoral catheter into the hepatic artery. Following treatment with SIR-Spheres, patients took 160 mg regorafenib orally once daily on Days 1-21 of each 28-day treatment cycle
Period: Overall Study
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
Started | 25 | 1
Completed | 0 | 0
Not Completed | 25 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Progressive Disease | 18 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib | Total
Number analyzed (Participants) | 25 | 1 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 1 | 18
  >=65 years | 8 | 0 | 8
Age, Continuous [Median (Full Range); unit: years] | 56 [44 to 79] | 64 [64 to 64] | 56 [44 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 0 | 13
  Male | 12 | 1 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 22 | 1 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 1 | 26

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Treatment-Related Adverse Events and Serious Adverse Events as a Measure of Safety
Description: A treatment-related adverse event or serious adverse event was any untoward medical occurrence in a participant which was considered to have a relationship with the study drug (suspected to be possibly or probably related to the study drug per the Investigator's assessment). Adverse events and serious adverse events will be assessed according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V4.03.
Time Frame: up to 15 months
Population: All patients who receive at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
Number analyzed (Participants) | 25 | 1
Participants | 25 | 1

2. Secondary Outcome: Number of Patients With an Objective Response (CR or PR)
Description: Defined as the number of patients with objective evidence of complete or partial response (CR or PR) using RECIST v 1.1. A CR is the complete disappearance of all target lesions. A PR is a decrease in of 30% or more of the diameter(s) of all target lesions from the baseline sum of diameters.
Time Frame: At 6 and 12 weeks after SIR-Spheres, and every 8 weeks thereafter, up to 18 months
Population: Includes all patients who have received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
Number analyzed (Participants) | 25 | 1
Participants | 1 | 0

3. Secondary Outcome: Median Progression-Free Survival
Description: Defined as the time (in months) from date of randomization to the date of first observation of progression based on radiological assessment by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1, or date of death from any cause, in the absence of progressive disease (PD) or censored at the date of last adequate tumor assessment. Progressive Disease is defined by RECIST v1.1 as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum while on study (this includes the baseline sum if that is the smallest on study), or the appearance of one or more new lesions.
Time Frame: At 6 and 12 weeks after SIR-Spheres, and every 8 weeks thereafter, up to 18 months.
Population: Includes all patients who received treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
Number analyzed (Participants) | 25 | 1
months | 3.7 [2.6 to 9.7] | NA [NA to NA] — Not reached at this time

4. Secondary Outcome: Median Overall Survival
Description: Defined as the time (in months) from date of randomization to date of death from any cause, or censored at the date last known alive.
Time Frame: up to 18 months
Population: Includes all patients who received treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
Number analyzed (Participants) | 25 | 1
Months | 12.1 [6.0 to 16.4] | NA [NA to NA] — Not reached at this time.

ADVERSE EVENTS:
Time Frame: Up to 15 months.
Description: All patients who received at least one dose of protocol treatment were followed for safety. Adverse events and serious adverse events were collected from day of first dose to 30 days after last protocol treatment and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Arm/Group | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib | Cohort 2: SIR-Spheres/Regorafenib
All-Cause Mortality (participants affected / at risk) | 16/25 | 0/1
Serious Adverse Events (participants affected / at risk) | 10/25 | 0/1
Other Adverse Events (participants affected / at risk) | 25/25 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib (N=25) | Cohort 2: SIR-Spheres/Regorafenib (N=1)
Constipation (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Regorafenib/SIR-Spheres/Regorafenib (N=25) | Cohort 2: SIR-Spheres/Regorafenib (N=1)
ANAEMIA (Blood and lymphatic system disorders) | 6 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0
MOTION SICKNESS (Ear and labyrinth disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 1
ASCITES (Gastrointestinal disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 9 | 1
DIARRHOEA (Gastrointestinal disorders) | 10 | 0
DRY MOUTH (Gastrointestinal disorders) | 3 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 1 | 0
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 | 0
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 | 0
GINGIVAL BLEEDING (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 11 | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1 | 0
ORAL PAIN (Gastrointestinal disorders) | 1 | 0
SENSITIVITY OF TEETH (Gastrointestinal disorders) | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 3 | 0
VOMITING (Gastrointestinal disorders) | 6 | 1
ASTHENIA (General disorders) | 4 | 0
CHILLS (General disorders) | 3 | 0
FATIGUE (General disorders) | 18 | 1
HERNIA (General disorders) | 1 | 0
HERNIA PAIN (General disorders) | 1 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0
MALAISE (General disorders) | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 5 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0
PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 4 | 0
SWELLING (General disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 1 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 1 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 0
NON-ALCOHOLIC STEATOHEPATITIS (Hepatobiliary disorders) | 1 | 0
PORTAL HYPERTENSION (Hepatobiliary disorders) | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 1 | 0
CANDIDA INFECTION (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 1 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0
SEPSIS (Infections and infestations) | 2 | 0
SKIN CANDIDA (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 4 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0
STOMA SITE IRRITATION (Injury, poisoning and procedural complications) | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 6 | 1
BLOOD ALBUMIN DECREASED (Investigations) | 1 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 | 0
BLOOD BILIRUBIN DECREASED (Investigations) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 7 | 0
BLOOD CALCIUM DECREASED (Investigations) | 1 | 0
BLOOD CHLORIDE DECREASED (Investigations) | 1 | 0
BLOOD CREATININE INCREASED (Investigations) | 2 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 | 0
BLOOD PHOSPHORUS DECREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
BLOOD SODIUM DECREASED (Investigations) | 1 | 0
CARCINOEMBRYONIC ANTIGEN INCREASED (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 | 0
PARACENTESIS (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 2 | 0
PLATELET COUNT INCREASED (Investigations) | 1 | 0
PROTEIN TOTAL DECREASED (Investigations) | 1 | 0
WEIGHT DECREASED (Investigations) | 3 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 12 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 2 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 5 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 | 0
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BALANCE DISORDER (Nervous system disorders) | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 5 | 0
HYPOAESTHESIA (Nervous system disorders) | 1 | 0
MIGRAINE (Nervous system disorders) | 1 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 | 0
SEIZURE (Nervous system disorders) | 1 | 0
TREMOR (Nervous system disorders) | 3 | 0
ABNORMAL DREAMS (Psychiatric disorders) | 1 | 0
ANXIETY (Psychiatric disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
DEPRESSION (Psychiatric disorders) | 2 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 1 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 1 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 1 | 0
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
VULVA CYST (Reproductive system and breast disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 6 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PARANASAL SINUS HYPERSECRETION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 6 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 2 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 4 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 3 | 0
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 2 | 0
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 | 0
CHEST TUBE INSERTION (Surgical and medical procedures) | 1 | 0
HERNIA REPAIR (Surgical and medical procedures) | 1 | 0
SKIN DISORDER NOT OTHERWISE SPECIFIED (Skin and subcutaneous tissue disorders) | 1 | 0
HOT FLUSH (Vascular disorders) | 1 | 0
HYPERTENSION (Vascular disorders) | 5 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 0
PERIPHERAL COLDNESS (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2014-04-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02195011/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT02195011/SAP_001.pdf